CLINICAL TRIAL: NCT05824546
Title: uSINE-PAMS Artificial Intelligence Driven, Ultrasound-Guided Lumbar Puncture to Improve Procedural Accuracy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Neuroscience Institute (Other)
Collaborators: HiCura Medical Pte Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: uSINE
Record Dates: First submitted 2023-03-22; First posted 2023-04-21 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-04

CONDITIONS: Ultrasound Therapy; Lumbar Puncture

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- uSINE-PAMS-guided (Experimental): Patients will undergo LP using uSINE-PAMS-guided technique
  Interventions: Procedure: Intervention Arm (uSINE-PAMS-technique)

INTERVENTIONS:
Procedure: Intervention Arm (uSINE-PAMS-technique) — Patients will be lying in a lateral recumbent position and in a fetal position with the neck, back and limbs held in flexion. L3-L4 inter-vertebral space will be identified by palpation of external landmarks of the patients' iliac crests and spinous process of lumbar vertebrae L3, L4 and L5 and confirmed using uSINE-integrated ultrasound. The angle of needle during needle advancement will also be determined using the uSINE-integrated ultrasound. Markings on the patients' skin surface will be made using PAMS (non-sterile component) to enable relocation of the site and angle of the needle entry. Patients' back will be cleaned and draped using aseptic technique. Next, local anaesthesia is infiltrated into the previously identified needle entry site before the LP needle is inserted with location and angulation according to PAMS (sterile component) guidance.

SUMMARY:
This study aims to test the effectiveness of uSINE-PAMS technology for lumbar puncture compared to traditional landmark-based technique. uSINE is a machine-learning software designed to aid the operators in ultrasound-guided lumbar puncture while PAMS is a two-part hardware to translate data from ultrasound to accurate needle insertion and angulation.

DETAILED DESCRIPTION:
Lumbar puncture (LP) is a routine invasive procedure performed for the diagnosis and treatment of central nervous system disorders. The traditional landmark-based method is associated with a high failure rate of up to 50%, leading to complications including back pain and epidural hematoma, diagnostic delay, and increased healthcare costs. The success rate has been improved with ultrasound guided LP but the use of ultrasound-guided LP has not been widespread due to inadequate training in ultrasound use and the inability to translate information derived from ultrasonography to the LP procedure. uSINE-PAMS was designed to address these challenges: uSINE is a machine-learning software to aid the operators in ultrasound-guided LP; PAMS is a two-part hardware to translate data from ultrasound to accurate needle insertion and angulation.

This study consists of a pilot phase to test the usability of uSINE-PAMs and allow for improvement in technology and clinical workflow for uSINE-PAMS. In the pilot phase, experienced NNI clinicians who have participated in a previous healthy volunteer study and have been trained to use uSINE will be the operators performing the uSINE-PAMS-guided lumbar puncture. During and upon completion of the study, challenges in the use of uSINE and PAMS to conduct LP as well as in the implementation of uSINE-PAMS in the clinical workflow will be determined and addressed prior to the main study, open-label single-arm phase 2 clinical trial. Ten patients will be recruited in this pilot phase.

Following the pilot phase, an open-label single-arm phase 2 clinical trial to test the effectiveness of uSINE-PAMS-guided LP against historical data of 55% from traditional landmark-based method. 50 patients who are planned for LP will be recruited to undergo LP using the uSINE-PAMS-guided technique. The overall hypothesis is that uSINE-PAMS-guided LP will achieve at least 20% improvement in first pass success rate of obtaining cerebrospinal fluid compared to historical data of 55% from traditional landmark-based technique, therefore leading to reduction in complication rates.

ELIGIBILITY:
INCLUSION CRITERIA:

* Patients planned for lumbar puncture as part of their clinical care
* 21 years of age or older
* Able to provide informed consent

EXCLUSION CRITERIA:

* Allergy to ultrasound gel
* Previous lumbar spinal instrumentation
* Patients with suspected spinal epidural abscess or any other infection at the potential site of needle entry on the back
* Possible raised intracranial pressure with risk of cerebral herniation, including presence of obstructive hydrocephalus, intracranial space-occupying lesion and cerebral edema
* Presence of significant thrombocytopenia (platelet <40k) or other bleeding diathesis; patients on antiplatelet and/or anticoagulation may be included if their antiplatelet and/or anticoagulation can be and are stopped for an adequate duration prior to lumbar puncture according to the institution guidelines.

Ages: 21 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-05-26 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
First pass success rate of obtaining CSF using uSINE-PAMS-guided technique against the traditional landmark-based method of 55%.technique against the traditional landmark-based method of 55%. | During procedure
  First pass is defined as the first LP attempt without withdrawing the LP needle out of the skin.

SECONDARY OUTCOMES:
Number of needle redirections using uSINE-PAMS-guided technique. | During procedure
  Needle redirection is defined as the number of times the LP needle was repositioned to obtain the CSF without withdrawing out of the skin.
Rate of traumatic LP using uSINE-PAMS-guided technique. | 1 hour after procedure
  Traumatic LP is defined as needle-induced blood (>5 red blood cells/ul) in the cerebrospinal fluid; Cases where red blood cells are expected in the cerebrospinal fluid will be excluded from this analysis.
Pain score from LP using uSINE-PAMS-guided technique. | Immediately after procedure
  Pain score will be assessed using the Universal Pain Assessment Tool which has a scale of 0-10, with 0 being no pain and 10 being Worst Pain Possible.
Rate of back pain that develops within 24 hours of the LP using uSINE-PAMS-guided technique. | Approximately 24 hours after procedure
  Pain score will be assessed using the Universal Pain Assessment Tool which has a scale of 0-10, with 0 being no pain and 10 being Worst Pain Possible.

OTHER OUTCOMES:
Rate of serious complications from LP using uSINE-PAMS-guided technique. | Within 1 week of procedure
  Serious complications include spinal hematoma, subdural hematoma, central nervous system infection and headaches requiring hospitalizations
Influence of BMI on the success or failure of the uSINE-PAMS-guided LP. | within 1 week of procedure

CONTACTS AND LOCATIONS:
Locations (1):
- National Neuroscience Institute (NNI), Singapore, Singapore

REFERENCES:
- [Derived] Lin X, Lam MLC, Chuang DF, Yuen JYE, Fu L, Jun Zhi Teh V, Marliya A, Saffari SE, Lim CSJ, Wong YL, Seet YHC. uSINE-PAMS Artificial Intelligence-Driven, Ultrasound-Guided Lumbar Puncture to Improve Procedural Accuracy: A Pilot Study Report. Neurol Clin Pract. 2025 Apr;15(2):e200447. doi: 10.1212/CPJ.0000000000200447. Epub 2025 Feb 25. PMID 40201070